CLINICAL TRIAL: NCT07076693
Title: Standard-of-care Systemic Therapy With or Without Local Therapy in Patients With Oligoprogressive NSCLC: A Prospective, Randomized Controlled Phase II/III Clinical Trial
Brief Title: Standard-of-care Systemic Therapy With or Without Local Therapy in Patients With Oligoprogressive Non-Small Cell Lung Cancer(NSCLC）
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xuwei Cai, Director, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IS25085
Record Dates: First submitted 2025-07-02; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: OligoProgressive Metastatic Disease; Non-Small Cell Lung Cancer
Keywords: oligopregressive disease; local therapy; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Parallel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): For patients with oligoprogressive disease, local treatment (radiotherapy or surgery) is administered to all/partial oligoprogressive sites while providing standard systemic therapy for 4-6 cycles. Radiotherapy is administered with radiation dose 30-50Gy. The site and regimen of radiotherapy or surgery are primarily determined by the investigator. Maintenance therapy or not is determined by investigator assessment after evaluation .
  Interventions: Procedure: Radiotherapy or Surgery; Drug: Standard Medical Therapy
- Active Comparator (Active Comparator): Standard systemic therapy is administered for 4-6 cycles. Maintenance therapy or not is determined by investigator assessment after evaluation.
  Interventions: Drug: Standard Medical Therapy

INTERVENTIONS:
Procedure: Radiotherapy or Surgery — Metastatic lesions were treated with surgical resection or radiotherapy. Surgical duration was determined by investigator assessment and metastatic or primary lesions were resected with palliative intent. Radiation dose and fractionation are 30~50Gy. Radiation dose, fractionation regimen, and treatment sites for metastatic lesions were determined at the investigator's discretion based on clinical indications.
  Arms: Experimental
Drug: Standard Medical Therapy — Patients with squamous cell carcinoma received docetaxel administered in 3-week cycles, and patients with adenocarcinoma received pemetrexed, patinum and one of sintilimab or ivonescimab.

SUMMARY:
This is a randomized, controlled, phase II/III clinical study to evaluate the efficacy and safety of stand-of-care systemic therapy with local therapy versus stand-of-care systemic therapy in patients with oligoprogressive non-small cell lung cancer(NSCLC).

DETAILED DESCRIPTION:
Subjects who meet all the inclusion criteria but do not meet any exclusion criteria are randomized into two groups at a ratio of 1:1: according to the stratification factors as below:

* mutation status (known vs absent/unknown)
* Number of oligoprogressive lesions (1-2 vs 3) Experimental group: For patients with oligoprogressive disease, local treatment (radiotherapy or surgery) is administered to all/partial oligoprogressive sites while providing standard systemic therapy for 4-6 cycles. Radiotherapy is administered with radiation dose 30-50Gy. The site and regimen of radiotherapy or surgery are primarily determined by the investigator. Maintenance therapy is determined by investigator assessment after evaluation.

Control group: Standard systemic therapy is administered for 4-6 cycles . Maintenance therapy is determined by investigator assessment after evaluation.

Adverse events (AEs) will be monitored throughout the study, and the severity will be graded to the guidelines listed in National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) version 5.0 or above. The safety will be followed up in the subjects who have received study treatment and discontinued the drug prematurely. All the subjects will be followed up for overall survival, until death, withdrawal of informed consent or end of study.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent form and voluntarily participate in this study;
2. Age 18-75 years;
3. ECOG 0-1, or able to tolerate radiotherapy/surgery and subsequent systemic therapy;
4. For Epidermal Growth Factor Receptor (EGFR)-sensitive mutant non-squamous NSCLC patients, first-line treatment must be the third-generation TKIs or progression after first/second-generation TKI without harboring T790M mutation, with ≤3 progressive lesions and ≤3 metastatic organs (PET-CT + cranial MRI preferred, or comprehensive imaging assessment, pathological examination not mandatory);
5. For squamous cell lung cancer patients, progression after first-line immunotherapy/chemotherapy-immunotherapy with ≤3 progressing lesions and ≤3 metastatic organs (PET-CT + cranial MRI preferred, or comprehensive imaging assessment, pathological examination not mandatory);
6. Expected survival ≥6 months;
7. No severe medical conditions;
8. Normal major organ functions, including:

   1. Blood tests: WBC count ≥4.0×10⁹/L, neutrophil count ≥1.5×10⁹/L, platelet count ≥80×10⁹/L, hemoglobin ≥90 g/L;
   2. Blood biochemistry: total bilirubin ≤1.5×ULN, ALT ≤2.5×ULN, AST ≤2.5×ULN, serum creatinine ≤1.5×ULN, or creatinine clearance ≥50 mL/min;
   3. Coagulation function: INR ≤1.5×ULN; APTT ≤1.5×ULN; FEV1 > 0.75 L;
9. All oligoprogressive sites must be tolerable for radiotherapy or surgical treatment; for patients receiving radiotherapy, if prior radiotherapy was administered to the primary lesion, the re-irradiated site must be the metastatic lesions;
10. No other primary tumors before treatment;
11. PD-L1 expression status and driver gene sensitive mutations are both acceptable;
12. At least one evaluable target lesion, with metastases occurring within one month defined as synchronous metastases;
13. Patients may have more than 3 metastatic sites in total with only 1-3 progressive lesions and no more than 3 metastatic organs (RECIST criteria; mediastinal lymph nodes and primary lesions not counted in the oligopregressive lesions);
14. For patients with treated CNS disease, eligibility requires stable brain metastases on imaging and clinically, no evidence of cavitation or hemorrhage in brain lesions, asymptomatic status, and no need for steroids (must discontinue steroids at least 1 week before randomization); symptomatic brain metastases, multiple brain metastases, or other emergencies may receive palliative treatment before randomization (at least 1 week).

Exclusion Criteria:

1. Large cell neuroendocrine carcinoma, pulmonary carcinoid tumor, or mixed small cell and small cell lung cancer;
2. Patients with progressive lesions over 3 lesions;
3. Patients with meningeal metastasis, pleural metastasis, or severe pleural/ascitic effusion, or those who had severe pleural effusion during prior treatment but are now controlled;
4. Patients with any other current or previous malignancies, except for non-melanoma skin cancer or carcinoma in situ of the cervix;
5. Any other disease or condition that contraindicates radiotherapy/chemotherapy/immunotherapy (e.g., active infection, within 6 months after myocardial infarction, symptomatic heart disease including unstable angina, congestive heart failure, or uncontrolled arrhythmia, immunosuppressive therapy);
6. Other conditions deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 7 weeks after standard subsequent-line therapy
  The proportion of patients achieving complete remission (CR) or partial remission (PR)
Progression-free survival (PFS) | up to 3 years
  Time from randomization to disease progression or death

SECONDARY OUTCOMES:
Overall survival (OS) | up to 3 years
  The time from random entry to death for any cause
Local Control (LC) | up to 3 years
  The time from the start of radiotherapy to any objectively recorded tumor progression at the irradiated site
Adverse Events (AE) | up to 3 years
  Number of participants with adverse events as assessed by CTCAE v5.0
local treatment tolerability | up to 3 years
  Number of participants with severe treatment--related adverse events as assessed by CTCAE v5.0 or who discontinue treatment
treatment failure pattern | up to 3 years
  The sites of disease progression post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Recruiting, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
yes
Supporting Information: Study Protocol